CLINICAL TRIAL: NCT06526962
Title: Comparison Between Two Different Tools for Outpatient Hysteroscopic Polypectomy: 5Fr Bipolar Electrode vs. Conical Optical 5Fr Fibers for Dual Wave-length Diode Laser
Brief Title: 5Fr Bipolar Electrode vs. Conical Optical 5Fr Fibers for Dual Wave-length Diode Laser for Hysteroscopic Polypectomy
Acronym: HYSTOP
Status: Recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Salvatore Giovanni Vitale, Professor, University of Cagliari
Other Study IDs: HYSTOP
Record Dates: First submitted 2024-07-16; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Endometrial Polyp
Keywords: Hysteroscopy; Outpatient; Endometrial Polyp; Polypectomy; Dual Wave-Lenght Diode Laser

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Endometrial Polyp
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients who undergo outpatient hysteroscopic polypectomy using 5Fr bipolar electrode
  Interventions: Device: 5Fr hysteroscopic bipolar electrode or conical optical 5Fr fibers for dual wave-length diode laser
- Group B: Patients who undergo outpatient hysteroscopic polypectomy using a conical optical 5Fr fibers for dual wave-length diode laser
  Interventions: Device: 5Fr hysteroscopic bipolar electrode or conical optical 5Fr fibers for dual wave-length diode laser

INTERVENTIONS:
Device: 5Fr hysteroscopic bipolar electrode or conical optical 5Fr fibers for dual wave-length diode laser — Outpatient hysteroscopic polypectomy

SUMMARY:
The primary objective of this study is to compare the performance of two different surgical instruments, the 5 Fr bipolar electrode and the 5 Fr angled conical optical fiber for dual wavelength diode laser, in performing hysteroscopic polypectomy in an outpatient setting.

DETAILED DESCRIPTION:
More specifically, the study aims to compare these instruments by evaluating the following parameters:

* Duration of the procedure;
* Use of any additional accessory instrumentation;
* Effectiveness of the procedure;
* Safety of the procedure;
* Adequacy of the operative specimen for histological analysis;
* Overall suitability of the instrument used;
* Levels of pain and anxiety perceived by the patient during the procedure;
* Changes in the patient's quality of life related to the persistence or resolution of symptoms following the procedure.

A prospective observational study will be conducted at the Obstetrics and Gynecology Clinic of the University Hospital "Duilio Casula" in Monserrato (Italy), following the approval of the study design by the Ethics Committee. Women who meet the inclusion and exclusion criteria will undergo a thorough medical history and gynecological clinical evaluation before performing diagnostic and operative hysteroscopy (T0). The characteristics of the participants, including age, ethnicity, weight, height, lifestyle habits, and medication use, will be recorded in a dedicated database. Each patient will be assigned an ID, which will serve as the patient's unique identifier.

Before performing the hysteroscopic procedure, each patient recruited for the study (T0) will undergo a thorough pelvic ultrasound evaluation using a transvaginal probe by an experienced sonographer (at least 500 procedures performed) according to standard protocols to evaluate the ultrasonographic characteristics of the endometrial polyp. Specifically, the location, size, echostructure, and vascular pattern will be carefully assessed and recorded. During the recruitment phase (T0), the EuroQol-5D questionnaire will be administered to determine the impact of symptoms related to the presence of the lesion on the patient's perceived quality of life. The Italian version of the EuroQol-5D questionnaire, validated by the EuroQoL Group, will be used for this study.

All recruited patients will then undergo diagnostic and operative hysteroscopy (T1) in an outpatient setting without any anesthesia/sedation or pharmacological/mechanical cervical preparation, using a 5 mm continuous flow Bettocchi rigid hysteroscope with a 5 Fr (1.67 mm) working channel and 30° optics (Karl Storz SE & Co. KG, Tuttlingen, Germany), performed by the same experienced operator (at least 500 procedures performed). The procedures will be carried out using a vaginoscopic approach. Uterine cavity distension will be achieved using saline solution, delivered by an electronic irrigation/aspiration pump (Endomat, Karl Storz SE & Co. KG, Tuttlingen, Germany), maintaining an intracavitary pressure ≤ 50 mmHg and an intrauterine flow ≤ 300 mL/min. Illumination will be provided by a 300 W Xenon light source. Images will be displayed on a high-resolution color monitor using an integrated circuit camera, and all procedures will be video recorded from the introduction of the hysteroscope until its extraction.

In this study phase, endocavitary characterization of endometrial polyps will be performed based on their size, location, and relationship to the tubal ostia, as well as their consistency and implantation base characteristics. Patients will then undergo polypectomy using one of two possible instruments: a 5 Fr "twizzle" bipolar electrode or a 5 Fr angled conical optical fiber for a dual-wavelength diode laser. The choice of instrument for each operative procedure will be at the operator's discretion.

During the procedure, the operator will be assisted by two assistants: one will manage the instrumentation, and the other will record the time required for the procedure and any use of additional accessory instrumentation, following the operator's instructions. Additionally, the latter will document on a dedicated form any events or symptoms experienced by the patient during the procedure and the 30-minute post-procedure observation period. The performance of each instrument will be subjectively evaluated by the operator regarding its cutting and coagulation precision, using a numerical rating scale from 0 to 10, where 0 indicates the minimum value and 10 the maximum value (Numerical Rating Scale, NRS). Furthermore, the adequacy of the removed sample for histological investigation will be assessed by the pathologist using a similar numerical rating scale (0 to 10, where 0 indicates the minimum appropriateness and 10 the maximum). Elements that may characterize the sample's adequacy include sufficient tissue quantity, absence of crushing, tearing, or electrocution artifacts, and adequate fixation.

Twenty minutes after completing the hysteroscopy (T2), the patient's perception of pain and anxiety levels experienced during the procedure will be assessed. The intensity of perceived pain will be evaluated using the VAS Scale (with levels ranging from 0 to 10, where 0 refers to no pain, 1-3 mild pain, 4-7 moderate pain, 8-10 severe pain) and the McGill Pain Questionnaire (which investigates perceived pain levels across three dimensions: sensory, affective, and evaluative). Anxiety levels experienced during the procedure will be assessed using the Hospital Anxiety and Depression Scale (H.A.D.S.). If the postoperative course is regular, patients will be discharged 30 minutes after the hysteroscopy.

Each patient will then undergo a post-surgical follow-up (T3) 60 days after the procedure, during which a thorough pelvic ultrasound evaluation will be performed (using the same previously described methods) primarily to investigate the possible presence of residual formations. The EuroQol-5D questionnaire will be administered again, and any late surgical complications will be recorded on a dedicated evaluation form.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years and < 60 years;
* suspicion of a single endometrial polyp, documented by ultrasound, with dimensions less than 20 mm;
* presence of abnormal uterine bleeding or history of infertility (defined as absence of conception after 12 months of regular unprotected intercourse aimed at conception);
* consent to participate in the study.

Exclusion Criteria:

* presence of multiple endometrial polyps;
* presence of a single endometrial polyp with dimensions greater than 20 mm;
* concurrent presence of intrauterine fibroids, focal or diffuse endometrial thickening, and/or intrauterine adhesions (synechiae);
* current or recent use (< 3 months) of anticoagulant drugs and/or Selective Estrogen Receptor Modulators (SERMs);
* presence of another known cause of vaginal/cervical bleeding;
* suspected adnexal pathology;
* confirmed diagnosis of endometrial cancer;
* suspected acute pelvic inflammation or recent history of pelvic inflammation (< 6 months);
* presence of tight cervical canal stenosis;
* requirement for any type of anesthesia to perform the hysteroscopic procedure.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with an indication for diagnostic and/or operative outpatient hysteroscopic polypectomy
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-11-07 (Estimated); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Time required to perform the operative hysteroscopic procedure. | End of procedure
  The time required to perform the operative hysteroscopic procedure, which will be measured in seconds from the entry into the uterine cavity until the completion of the procedure, defined as the complete resection of the lesion (excluding the time related to the extraction of the resected material).

SECONDARY OUTCOMES:
Need for supplementary instrumentation | End of procedure
  The need for supplementary instrumentation to complete the procedure (e.g., 5 Fr cold blade scissors)
Effectiveness in removing the lesions | 60 days
  Effectiveness of the procedure (absence/persistence of the lesion), documented by postoperative ultrasound evaluation performed 60 days after the procedure
Adverse events | 30 minutes
  Adverse events related to the procedure (e.g., vagal syndromes, bleeding, uterine perforations, or other injuries to the uterus and adjacent organs)
Quantity of resected tissue | 40 days
  Adequacy of the resected material weight for histological examination (weight in grams)
Instrument Suitability | End of procedure
  Overall suitability of the instrument used (in terms of its cutting and coagulation precision), as judged by the operating surgeon
Pain perception | 20 minutes
  The level of pain perceived by the patient during the procedure, evaluated using the Visual Analog Scale (VAS, from a minimum value of 1 to a maximum value of 10, where 1 is the best outcome and 10 is the worst outcome)
Level of anxiety during the procedure | 20 minutes
  Level of anxiety experienced by the patient during the procedure, evaluated using the Hospital Anxiety and Depression Scale (H.A.D.S.), from a minimum value of 0 to a maximum value of 21, where 0 is the best outcome and 21 is the worst outcome)
Patients' quality of life | 60 days
  Changes in the patient's perceived quality of life 60 days after the procedure, evaluated using the EuroQol-5D questionnaire (EuroQol 5-dimension questionnaire, from a minimum value of 0 to a maximum value of 100, where 0 is the worst outcome and 100 is the best outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salazar CA, Isaacson KB. Office Operative Hysteroscopy: An Update. J Minim Invasive Gynecol. 2018 Feb;25(2):199-208. doi: 10.1016/j.jmig.2017.08.009. Epub 2017 Aug 10. PMID 28803811
- [Background] Luerti M, Vitagliano A, Di Spiezio Sardo A, Angioni S, Garuti G, De Angelis C; Italian School of Minimally Invasive Gynecological Surgery Hysteroscopists Group. Effectiveness of Hysteroscopic Techniques for Endometrial Polyp Removal: The Italian Multicenter Trial. J Minim Invasive Gynecol. 2019 Sep-Oct;26(6):1169-1176. doi: 10.1016/j.jmig.2018.12.002. Epub 2018 Dec 7. PMID 30528831
- [Background] Vitale SG, Sapia F, Rapisarda AMC, Valenti G, Santangelo F, Rossetti D, Chiofalo B, Sarpietro G, La Rosa VL, Triolo O, Noventa M, Gizzo S, Lagana AS. Hysteroscopic Morcellation of Submucous Myomas: A Systematic Review. Biomed Res Int. 2017;2017:6848250. doi: 10.1155/2017/6848250. Epub 2017 Aug 29. PMID 28948169
- [Background] Bougie O, Lortie K, Shenassa H, Chen I, Singh SS. Treatment of Asherman's syndrome in an outpatient hysteroscopy setting. J Minim Invasive Gynecol. 2015 Mar-Apr;22(3):446-50. doi: 10.1016/j.jmig.2014.12.006. Epub 2014 Dec 10. PMID 25497164
- [Background] Bar-On S, Ben-David A, Rattan G, Grisaru D. Is outpatient hysteroscopy accurate for the diagnosis of endometrial pathology among perimenopausal and postmenopausal women? Menopause. 2018 Feb;25(2):160-164. doi: 10.1097/GME.0000000000000961. PMID 28763396
- [Background] Piecak K, Milart P. Hysteroscopic myomectomy. Prz Menopauzalny. 2017 Dec;16(4):126-128. doi: 10.5114/pm.2017.72757. Epub 2017 Dec 30. PMID 29483854
- [Background] Lasmar RB, Barrozo PR, Dias R, Oliveira MA. Submucous myomas: a new presurgical classification to evaluate the viability of hysteroscopic surgical treatment--preliminary report. J Minim Invasive Gynecol. 2005 Jul-Aug;12(4):308-11. doi: 10.1016/j.jmig.2005.05.014. PMID 16036188
- [Background] Lasmar RB, Xinmei Z, Indman PD, Celeste RK, Di Spiezio Sardo A. Feasibility of a new system of classification of submucous myomas: a multicenter study. Fertil Steril. 2011 May;95(6):2073-7. doi: 10.1016/j.fertnstert.2011.01.147. Epub 2011 Feb 21. PMID 21333985
- [Background] Lara-Dominguez MD, Arjona-Berral JE, Dios-Palomares R, Castelo-Branco C. Outpatient hysteroscopic polypectomy: bipolar energy system (Versapoint(R)) versus diode laser - randomized clinical trial. Gynecol Endocrinol. 2016;32(3):196-200. doi: 10.3109/09513590.2015.1105209. Epub 2015 Nov 3. PMID 26527251
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Van Den Bosch T, Verbakel JY, Valentin L, Wynants L, De Cock B, Pascual MA, Leone FPG, Sladkevicius P, Alcazar JL, Votino A, Fruscio R, Lanzani C, Van Holsbeke C, Rossi A, Jokubkiene L, Kudla M, Jakab A, Domali E, Epstein E, Van Pachterbeke C, Bourne T, Van Calster B, Timmerman D. Typical ultrasound features of various endometrial pathologies described using International Endometrial Tumor Analysis (IETA) terminology in women with abnormal uterine bleeding. Ultrasound Obstet Gynecol. 2021 Jan;57(1):164-172. doi: 10.1002/uog.22109. PMID 32484286
- [Background] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767